CLINICAL TRIAL: NCT03843632
Title: An Open-Label, Multicenter, Single-arm Study to Evaluate the Immunogenicity of VARIVAX™ in Healthy Russian Individuals 12 Months of Age and Older
Brief Title: Evaluation of the Immunogenicity and Safety of VARIVAX™ in Healthy Russians (V210-058)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V210-058; V210-058 (Other: Merck Protocol Number); 2019-003903-36 (EudraCT Number)
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Results first posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Varicella
MeSH Terms: conditions — Chickenpox | interventions — Chickenpox Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- VARIVAX™ (Experimental): All participants will receive one dose subcutaneous (SC) VARIVAX™ on Day 1. Adult participants and adolescent participants 13 years and older will also receive a second SC dose VARIVAX™ on Day 43.
  Interventions: Biological: VARIVAX™

INTERVENTIONS:
Biological: VARIVAX™ — VARIVAX™ administered by SC injection as 0.5 mL Varicella Virus Vaccine Live in sterile suspension on Day 1 (all participants) and Day 43 (adult and adolescent participants).

SUMMARY:
The purpose of this study was to evaluate the immunogenicity and safety of VARIVAX™ vaccine in healthy Russian children, adolescents, and adults. No formal hypothesis was tested.

ELIGIBILITY:
Inclusion Criteria:

* has a negative clinical history for varicella and herpes zoster
* females of reproductive potential have a negative pregnancy test prior to each study vaccination
* females of reproductive potential remain abstinent or use 2 acceptable methods of birth control during study until 3 months following last study vaccination
* females not of reproductive potential do not require a pregnancy test or use of contraceptives
* legal representative of adult or parent of children understands risks involved with, consent to participate in, and comply with the study procedures

Exclusion Criteria:

* has a history of allergy or anaphylactic reaction to neomycin, gelatin, or any component of VARIVAX^TM
* has received any form of varicella or herpes zoster vaccine at any time prior to study, or anticipates receiving any during study
* has received immune globulin, a blood transfusion or blood derived products within prior 5 months or plans to do so during study
* has received aspirin or any aspirin-containing products within prior 14 days
* has been exposed to varicella or herpes zoster in the prior 4 weeks involving playmate, hospital or continuous household contact, or had contact with a newborn whose mother had chickenpox 5 days before or 2 days after delivery
* has, or lives with a person who has, any congenital or acquired immune deficiency, neoplastic disease, or depressed immunity including those resulting from corticosteroid use or other immunosuppressive therapy
* has received glucocorticosteroids for more than 5 consecutive days within prior 3 months, or any dose of glucocorticoids within prior 7 days, or expects to use glucocorticosteroids during the study
* was vaccinated with licensed non-live or live vaccine within prior 30 days or expects vaccination during 42 day follow-up postvaccination period
* had a fever within 72 hours prior to study vaccination
* has participated in another trial within prior 30 days, is currently participating in another trial, or plans to participate in another trial during the planned study period for this trial
* is pregnant or nursing

Ages: 12 Months to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-06-19 (Actual); Study Completion 2020-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (5):
- Russia (5):
  - Republican Clinical Infectious Hospital n.a. A.F. Agafonov ( Site 5816), Kazan'
  - Research Institute of Children Infections ( Site 5801), Saint Petersburg
  - SPb Pasteur RI of Epidemiology and Microbiology ( Site 5817), Saint Petersburg
  - Smolensk State Medical University ( Site 5814), Smolensk
  - Smolensk State Medical University ( Site 5815), Smolensk

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Paradis EM, Tikhonov O, Cao X, Kharit SM, Fokin A, Platt HL, Wittke F, Jotterand V. Phase 3, open-label, Russian, multicenter, single-arm trial to evaluate the immunogenicity of varicella vaccine (VARIVAX) in healthy infants, children, and adolescents. Hum Vaccin Immunother. 2021 Nov 2;17(11):4183-4189. doi: 10.1080/21645515.2021.1975451. Epub 2021 Oct 26. PMID 34702124
- [Derived] Paradis EM, Tikhonov O, Cao X, Kharit SM, Fokin A, Platt HL, Banniettis N. Phase 3, open-label, Russian, multicenter, single-arm trial to evaluate the immunogenicity of varicella vaccine (VARIVAX) in healthy adults. Hum Vaccin Immunother. 2021 Nov 2;17(11):4177-4182. doi: 10.1080/21645515.2021.1957414. Epub 2021 Sep 2. PMID 34473594

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled healthy Russians aged 12 months and older. Additional inclusion criteria applied.
Pre-assignment Details: 150 participants were enrolled and received VARIVAX™ on study. Adults and Adolescents received 2 vaccinations on study and children received 1 vaccination.
Groups:
- VARIVAX Adults (18 to 75 Years): Participants aged 18 to 75 years of age received 2 doses of VARIVAX™ administered approximately six weeks apart: one 0.5 mL dose of VARIVAX™ administered by subcutaneous (SC) injection on Day 1, and a second 0.5 mL dose of VARIVAX™ by SC injection on Day 43.
- VARIVAX™ Adolescents 13 to 17 Years of Age: Participants aged 13 to 17 years of age received 2 doses of VARIVAX™ administered approximately six weeks apart: one 0.5 mL dose of VARIVAX™ administered by SC injection on Day 1, and a second 0.5 mL dose of VARIVAX™ by SC injection on Day 43.
- VARIVAX™ Children 7 to 12 Years of Age: Participants aged 7 to 12 years of age received one 0.5 mL dose of VARIVAX™ administered by SC injection on Day 1.
- VARIVAX™ Children 12 Months to 6 Years of Age: Participants aged 12 months to 6 years of age received one 0.5 mL dose of VARIVAX™ administered by SC injection on Day 1.
Period: Overall Study
Arm/Group | VARIVAX Adults (18 to 75 Years) | VARIVAX™ Adolescents 13 to 17 Years of Age | VARIVAX™ Children 7 to 12 Years of Age | VARIVAX™ Children 12 Months to 6 Years of Age
Started | 50 | 30 | 33 | 37
Vaccination 1 | 50 | 30 | 33 | 37
Vaccination 2 | 49 | 30 | 0 | 0
Completed | 49 | 30 | 33 | 37
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VARIVAX Adults (18 to 75 Years) | VARIVAX™ Adolescents 13 to 17 Years of Age | VARIVAX™ Children 7 to 12 Years of Age | VARIVAX™ Children 12 Months to 6 Years of Age | Total
Number analyzed (Participants) | 50 | 30 | 33 | 37 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.7 (6.0) | 15.1 (1.5) | 9.6 (1.6) | 3.2 (1.6) | 14.2 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 16 | 14 | 18 | 84
  Male | 14 | 14 | 19 | 19 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 48 | 30 | 33 | 37 | 148
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 50 | 30 | 33 | 37 | 150
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Serostatus for Varicella-Zoster Virus (VZV) [Count of Participants; unit: Participants] — VZV seronegative status at baseline was VZV antibody titer <1.25 glycoprotein enzyme-linked immunosorbent assay (gpELISA) units/mL at baseline. A VZV seropositive status at baseline was a VZV antibody titer ≥1.25 gpELISA units/mL).
  Participants
    VZV Seronegative | 26 | 18 | 22 | 34 | 100
    VZV Seropositive | 24 | 12 | 11 | 3 | 50

OUTCOME MEASURES:

1. Primary Outcome: Varicella Zoster Virus (VZV) Antibody Response Rate at 6 Weeks Post Last Vaccination in Participants Who Were Seronegative at Baseline
Description: VZV antibody titers were measured using a glycoprotein enzyme-linked immunosorbent assay (gpELISA). The VZV antibody response rate was defined as the percentage of participants with a post-vaccination VZV antibody titer ≥5 gpELISA units/mL for participants whose baseline VZV antibody titer was <1.25 gpELISA units/mL. VZV antibody response rate was reported for all study arms at 6 weeks post last vaccination (Vaccination 1 for children and Vaccination 2 for adults and adolescents) for participants who were seronegative to VZW at baseline.
Time Frame: Adults and Adolescents: 6 weeks post Vaccination 2 (up to approximately 86 days), Children: 6 weeks post Vaccination 1 (up to approximately 43 days)
Population: All allocated participants without deviations from the protocol that would substantially affect the results of the immunogenicity outcome measures (Per-Protocol population) who were seronegative at baseline and who received Vaccination 1 (children) or Vaccination 1 and Vaccination 2 (adults and adolescents) were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | VARIVAX Adults (18 to 75 Years) | VARIVAX™ Adolescents 13 to 17 Years of Age | VARIVAX™ Children 7 to 12 Years of Age | VARIVAX™ Children 12 Months to 6 Years of Age
Number analyzed (Participants) | 26 | 18 | 22 | 34
Percentage of participants | 100.0 [86.8 to 100.0] | 100.0 [81.5 to 100.0] | 95.5 [77.2 to 99.9] | 100.0 [89.7 to 100.0]

2. Primary Outcome: Geometric Mean Titers (GMTs) of VZV Antibodies at 6 Weeks Post Last Vaccination in Participants Who Were Seronegative at Baseline
Description: GMTs of VZV antibodies were measured post-vaccination using a gpELISA. GMT was calculated at each time point by taking the log of the titers, averaging over all participants values, and then back-transforming to the original scale. GMT was reported for all study arms at 6 weeks post last vaccination (Vaccination 1 for children and Vaccination 2 for adults and adolescents) for participants who were seronegative to VZW at baseline.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | VARIVAX Adults (18 to 75 Years) | VARIVAX™ Adolescents 13 to 17 Years of Age | VARIVAX™ Children 7 to 12 Years of Age | VARIVAX™ Children 12 Months to 6 Years of Age
Number analyzed (Participants) | 26 | 18 | 22 | 34
gpELISA units/mL | 70.7 (47.9) [47.9 to 104.2] | 78.6 (46.5) [46.5 to 133.0] | 11.3 (7.3) [7.3 to 17.5] | 13.9 (11.2) [11.2 to 17.2]

3. Primary Outcome: VZV Antibody Seroconversion Rate at 6 Weeks Post Last Vaccination in Participants Who Were Seronegative at Baseline
Description: VZV antibody levels were measured using a gpELISA. The VZW antibody seroconversion rate was defined as the percentage of participants with VZV antibodies ≥1.25 gpELISA units/mL in participants with a baseline VZV antibody titer <1.25 gpELISA units/mL. VZW antibody seroconversion was reported for all study arms at 6 weeks post last vaccination (Vaccination 1 for children and Vaccination 2 for adults and adolescents) for participants who were seronegative to VZW at baseline.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | VARIVAX Adults (18 to 75 Years) | VARIVAX™ Adolescents 13 to 17 Years of Age | VARIVAX™ Children 7 to 12 Years of Age | VARIVAX™ Children 12 Months to 6 Years of Age
Number analyzed (Participants) | 26 | 18 | 22 | 34
Percentage of participants | 100.0 (86.8) [86.8 to 100.0] | 100.0 (81.5) [81.5 to 100.0] | 95.5 (77.2) [77.2 to 99.9] | 100.0 (89.7) [89.7 to 100.0]

4. Primary Outcome: GMTs of VZV Antibodies at Day 1 and 6 Weeks Post Last Vaccination in Participants Who Were Seropositive at Baseline
Description: GMTs of VZV antibodies were measured post-vaccination using a gpELISA. GMT was calculated at each time point by taking the log of the titers, averaging over all participants values, and then back-transforming to the original scale. GMT was reported for all study arms at 6 weeks post last vaccination (Vaccination 1 for children and Vaccination 2 for adults and adolescents) for participants who were seropositive to VZW at baseline. Per protocol, confidence intervals (CIs) were only calculated when there were at least 5 participants who were seropositive in a treatment group.
Time Frame: Day 1 (Baseline), 6 weeks post last vaccination (Day 43 for children and Day 84 for adults and adolescents)
Population: All allocated participants without deviations from the protocol that would substantially affect the results of the immunogenicity outcome measures (Per-Protocol population) who were seropositive at baseline and who received Vaccination 1 (children) or Vaccination 1 and Vaccination 2 (adults and adolescents) were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | VARIVAX Adults (18 to 75 Years) | VARIVAX™ Adolescents 13 to 17 Years of Age | VARIVAX™ Children 7 to 12 Years of Age | VARIVAX™ Children 12 Months to 6 Years of Age
Number analyzed (Participants) | 23 | 12 | 11 | 3
gpELISA units/mL
  Day 1 (Baseline) | 71.1 [31.4 to 161.2] | 13.4 [5.8 to 31.0] | 24.8 [7.2 to 85.5] | 4.2 [NA to NA] — Per protocol, CIs were not calculated when <5 participants were seropositive in a treatment group.
  Post Last Vaccination | 216.7 [132.8 to 353.6] | 151.7 [92.5 to 248.6] | 125.0 [37.9 to 411.7] | 47.6 [NA to NA] — Per protocol, CIs were not calculated when <5 participants were seropositive in a treatment group.

5. Primary Outcome: Geometric Mean Fold Rise (GMFR) in VZV Antibody Titers From Day 1 to 6 Weeks Post Last Vaccination in Participants Who Were Seropositive at Baseline
Description: GMTs were measured using a gpELISA. For participants who were seropositive at baseline (baseline VZV antibody titer ≥1.25 gpELISA units/mL), the GMFR was calculated as the ratio of the VZV GMT at 6 weeks post last vaccination to the VZV GMT at Day 1 (baseline). The GMFR from Day 1 was reported for all study arms at 6 weeks post last vaccination (Vaccination 1 for children and Vaccination 2 for adults and adolescents) for participants who were seropositive to VZW at baseline. Per protocol, CIs were only calculated when there were at least 5 participants who were seropositive in a treatment group.
Time Frame: Day 1 (Baseline), 6 weeks post last vaccination (Day 43 for children and Day 84 for adults and adolescents)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | VARIVAX Adults (18 to 75 Years) | VARIVAX™ Adolescents 13 to 17 Years of Age | VARIVAX™ Children 7 to 12 Years of Age | VARIVAX™ Children 12 Months to 6 Years of Age
Number analyzed (Participants) | 23 | 12 | 11 | 3
Ratio | 3.0 [2.0 to 4.8] | 11.3 [4.6 to 27.5] | 5.0 [2.6 to 9.7] | 11.2 [NA to NA] — Per protocol, CIs were not calculated when <5 participants were seropositive in a treatment group.

6. Primary Outcome: Percentage of Participants With ≥4-Fold Rise in Antibody Titers From Day 1 to 6 Weeks Post Last Vaccination Among Participants Who Were Seropositive at Baseline
Description: GMTs were measured using a gpELISA. For participants who were seropositive at baseline (baseline VZV antibody titer ≥1.25 gpELISA units/mL), the percentage of participants with a ≥4-fold rise in VZV antibody titer from Day 1 (baseline) to post-vaccination was assessed and reported for all study arms at 6 weeks post last vaccination (Vaccination 1 for children and Vaccination 2 for adults and adolescents). Per protocol, CIs were only calculated when there were at least 5 participants who were seropositive in a treatment group.
Time Frame: Day 1 (Baseline), 6 weeks post last vaccination (Day 43 for children and Day 84 for adults and adolescents)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | VARIVAX Adults (18 to 75 Years) | VARIVAX™ Adolescents 13 to 17 Years of Age | VARIVAX™ Children 7 to 12 Years of Age | VARIVAX™ Children 12 Months to 6 Years of Age
Number analyzed (Participants) | 23 | 12 | 11 | 3
Percentage of participants | 60.9 [38.5 to 80.3] | 66.7 [34.9 to 90.1] | 54.5 [23.4 to 83.3] | 100.0 [NA to NA] — Per protocol, CIs were not calculated when <5 participants were seropositive in a treatment group.

7. Secondary Outcome: Percentage of Participants With Solicited Injection-Site Adverse Events (AEs) Post-Vaccination 1
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited injection-site AEs, which included erythema, pain, and swelling, were recorded on a Vaccine Report Card (VRC). The percentage of participants who experienced solicited injection-site AEs after Vaccination 1 (up to approximately 5 days post-vaccination) was summarized for all study arms.
Time Frame: Up to approximately 5 days post-Vaccination 1
Population: All allocated participants who received at least one dose of study vaccine and who had some safety follow-up data after the respective vaccination were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | VARIVAX Adults (18 to 75 Years) | VARIVAX™ Adolescents 13 to 17 Years of Age | VARIVAX™ Children 7 to 12 Years of Age | VARIVAX™ Children 12 Months to 6 Years of Age
Number analyzed (Participants) | 50 | 30 | 33 | 37
Percentage of participants
  Injection-site erythema | 16.0 | 3.3 | 3.0 | 0.0
  Injection-site pain | 40.0 | 23.3 | 30.3 | 13.5
  Injection-site swelling | 10.0 | 0.0 | 3.0 | 0.0

8. Secondary Outcome: Percentage of Participants With Solicited Injection-Site AEs Post-Vaccination 2
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited injection-site AEs, which included erythema, pain, and swelling, were recorded on a VRC. The percentage of participants who experienced solicited injection-site AEs after Vaccination 2 (up to approximately 5 days post-vaccination) was summarized for all study arms receiving a second vaccination (adults and adolescents).
Time Frame: Up to approximately 5 days post-Vaccination 2 (up to approximately 48 days)
Population: All allocated participants who received two doses of study vaccine (adults and adolescents) and who had some safety follow-up data after the respective vaccination were analyzed. Per protocol, the two children study arms did not receive a second vaccination and were excluded from this analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | VARIVAX Adults (18 to 75 Years) | VARIVAX™ Adolescents 13 to 17 Years of Age | VARIVAX™ Children 7 to 12 Years of Age | VARIVAX™ Children 12 Months to 6 Years of Age
Number analyzed (Participants) | 49 | 30 | 0 | 0
Percentage of participants
  Injection-site erythema | 18.4 | 0 |  |
  Injection-site pain | 49.0 | 23.3 |  |
  Injection-site swelling | 8.2 | 3.3 |  |

9. Secondary Outcome: Percentage of Participants With Unsolicited Injection-Site AEs Post-Vaccination 1
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Unsolicited injection-site AEs were recorded on a VRC. The percentage of participants who experienced unsolicited injection-site AEs after Vaccination 1 (up to approximately 42 days post-vaccination) was summarized for all study arms.
Time Frame: Up to approximately 42 days post-Vaccination 1
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | VARIVAX Adults (18 to 75 Years) | VARIVAX™ Adolescents 13 to 17 Years of Age | VARIVAX™ Children 7 to 12 Years of Age | VARIVAX™ Children 12 Months to 6 Years of Age
Number analyzed (Participants) | 50 | 30 | 33 | 37
Percentage of participants | 2.0 | 3.3 | 0.0 | 5.4

10. Secondary Outcome: Percentage of Participants With Unsolicited Injection-Site AEs Post-Vaccination 2
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Unsolicited injection-site AEs were recorded on a VRC. The percentage of participants who experienced unsolicited injection-site AEs after Vaccination 2 (up to approximately 42 days post-vaccination) was summarized for all study arms receiving a second vaccination (adults and adolescents).
Time Frame: Up to approximately 42 days post-Vaccination 2 (up to approximately 86 days)
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | VARIVAX Adults (18 to 75 Years) | VARIVAX™ Adolescents 13 to 17 Years of Age | VARIVAX™ Children 7 to 12 Years of Age | VARIVAX™ Children 12 Months to 6 Years of Age
Number analyzed (Participants) | 49 | 30 | 0 | 0
Percentage of participants | 0.0 | 0.0 |  |

11. Secondary Outcome: Percentage of Participants With Elevated Temperature Post-Vaccination 1
Description: The participant's temperature was taken in the evening after Vaccination 1 and daily through Day 28, and was recorded on a VRC. An elevated temperature was defined as ≥39.0 °C (102.2 °F). The percentage of participants with elevated temperature after Vaccination 1 (up to approximately 28 days post-vaccination) was summarized for all study arms.
Time Frame: Up to 28 days post-Vaccination 1
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | VARIVAX Adults (18 to 75 Years) | VARIVAX™ Adolescents 13 to 17 Years of Age | VARIVAX™ Children 7 to 12 Years of Age | VARIVAX™ Children 12 Months to 6 Years of Age
Number analyzed (Participants) | 50 | 30 | 33 | 37
Percentage of participants | 2.0 | 0.0 | 3.0 | 8.1

12. Secondary Outcome: Percentage of Participants With Elevated Temperature Post-Vaccination 2
Description: The participant's temperature was taken in the evening after Vaccination 2 and daily through Day 28, and was recorded on a VRC. An elevated temperature was defined as ≥39.0 °C (102.2 °F). The percentage of participants with elevated temperature after Vaccination 2 (up to approximately 28 days post-vaccination) was summarized for all study arms receiving a second vaccination (adults and adolescents).
Time Frame: Up to 28 days post-Vaccination 2 (up to approximately 71 days)
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | VARIVAX Adults (18 to 75 Years) | VARIVAX™ Adolescents 13 to 17 Years of Age | VARIVAX™ Children 7 to 12 Years of Age | VARIVAX™ Children 12 Months to 6 Years of Age
Number analyzed (Participants) | 49 | 30 | 0 | 0
Percentage of participants | 0.0 | 0.0 |  |

13. Secondary Outcome: Percentage of Participants With Varicella- and Herpes Zoster-Like Rashes Post-Vaccination 1
Description: The development of varicella-like and herpes zoster-like rashes was recorded on a VRC. The percentage of participants who experienced varicella-like and herpes zoster-like rashes after Vaccination 1 (up to approximately 42 days post-vaccination) was summarized for all study arms.
Time Frame: Up to approximately 42 days post-Vaccination 1
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | VARIVAX Adults (18 to 75 Years) | VARIVAX™ Adolescents 13 to 17 Years of Age | VARIVAX™ Children 7 to 12 Years of Age | VARIVAX™ Children 12 Months to 6 Years of Age
Number analyzed (Participants) | 50 | 30 | 33 | 37
Percentage of participants
  Varicella-like rash | 6.0 | 0.0 | 6.1 | 2.7
  Herpes zoster-like rash | 0.0 | 0.0 | 0.0 | 0.0

14. Secondary Outcome: Percentage of Participants With Varicella- and Herpes Zoster-Like Rashes Post-Vaccination 2
Description: The development of varicella-like and herpes zoster-like rashes was recorded on a VRC. The percentage of participants who experienced varicella-like and herpes zoster-like rashes after Vaccination 2 (up to approximately 42 days post-vaccination) was summarized for all study arms receiving a second vaccination (adults and adolescents).
Time Frame: Up to approximately 42 days post-Vaccination 2 (up to approximately 86 days)
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | VARIVAX Adults (18 to 75 Years) | VARIVAX™ Adolescents 13 to 17 Years of Age | VARIVAX™ Children 7 to 12 Years of Age | VARIVAX™ Children 12 Months to 6 Years of Age
Number analyzed (Participants) | 49 | 30 | 0 | 0
Percentage of participants | 2.0 | 0.0 |  |

15. Secondary Outcome: Percentage of Participants With Systemic AEs Post-Vaccination 1
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A systemic AE was defined as any non-injection-site AE. Systemic AEs were recorded on a VRC. The percentage of participants who experienced a systemic AE after Vaccination 1 (up to approximately 42 days post-vaccination) was summarized for all study arms.
Time Frame: Up to approximately 42 days post-Vaccination 1
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | VARIVAX Adults (18 to 75 Years) | VARIVAX™ Adolescents 13 to 17 Years of Age | VARIVAX™ Children 7 to 12 Years of Age | VARIVAX™ Children 12 Months to 6 Years of Age
Number analyzed (Participants) | 50 | 30 | 33 | 37
Percentage of participants | 38.0 | 23.3 | 36.4 | 43.2

16. Secondary Outcome: Percentage of Participants With Systemic AEs Post-Vaccination 2
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A systemic AE was defined as any non-injection-site AE. Systemic AEs were recorded on a VRC. The percentage of participants who experienced a systemic AE after Vaccination 2 (up to approximately 42 days post-vaccination) was summarized for all study arms receiving a second vaccination (adults and adolescents).
Time Frame: Up to approximately 42 days post-Vaccination 2 (up to approximately 86 days)
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | VARIVAX Adults (18 to 75 Years) | VARIVAX™ Adolescents 13 to 17 Years of Age | VARIVAX™ Children 7 to 12 Years of Age | VARIVAX™ Children 12 Months to 6 Years of Age
Number analyzed (Participants) | 49 | 30 | 0 | 0
Percentage of participants | 28.6 | 26.7 |  |

17. Secondary Outcome: Percentage of Participants With 1 or More Serious Adverse Events (SAEs) Post-Vaccination 1 or Post-Vaccination 2
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was an AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or another important medical event. The percentage of participants who experienced one or more SAEs after either vaccination (up to approximately 42 days post-vaccination) was summarized for all study arms.
Time Frame: Up to 42 days post-Vaccination 1 or post-Vaccination 2 (up to approximately 86 days)
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | VARIVAX Adults (18 to 75 Years) | VARIVAX™ Adolescents 13 to 17 Years of Age | VARIVAX™ Children 7 to 12 Years of Age | VARIVAX™ Children 12 Months to 6 Years of Age
Number analyzed (Participants) | 50 | 30 | 33 | 37
Percentage of participants | 0.0 | 0.0 | 3.0 | 0.0

18. Secondary Outcome: Percentage of Participants With Vaccine-Related SAEs Post-Vaccination 1 or Post-Vaccination 2
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A vaccine-related SAE was an AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or another important medical event, that was considered at least possibly related to the study vaccine. The percentage of participants who experienced one or more vaccine-related SAEs after either vaccination (up to approximately 42 days post-vaccination) was summarized for all study arms.
Time Frame: Up to 42 days post-Vaccination 1 or post-Vaccination 2 (up to approximately 86 days)
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | VARIVAX Adults (18 to 75 Years) | VARIVAX™ Adolescents 13 to 17 Years of Age | VARIVAX™ Children 7 to 12 Years of Age | VARIVAX™ Children 12 Months to 6 Years of Age
Number analyzed (Participants) | 50 | 30 | 33 | 37
Percentage of participants | 0.0 | 0.0 | 0.0 | 0.0

19. Secondary Outcome: Percentage of Participants With Vaccine-Related Death Post-Vaccination 1 or Post-Vaccination 2
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A vaccine-related SAE was an AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or another important medical event, that was considered at least possibly related to the study vaccine. The percentage of participants who experienced a vaccine-related SAE that resulted in death after either vaccination (up to approximately 42 days post-vaccination) was summarized for all study arms.
Time Frame: Up to 42 days post-Vaccination 1 or post-Vaccination 2 (up to approximately 86 days)
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | VARIVAX Adults (18 to 75 Years) | VARIVAX™ Adolescents 13 to 17 Years of Age | VARIVAX™ Children 7 to 12 Years of Age | VARIVAX™ Children 12 Months to 6 Years of Age
Number analyzed (Participants) | 50 | 30 | 33 | 37
Percentage of participants | 0.0 | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Adverse Events: Up to 42 days post-Vaccination 1 or post-Vaccination 2 (up to approximately 86 days); All-Cause Mortality: Up to approximately 16 months
Description: All-Cause Mortality, Serious adverse events (AEs), and Other AE tables include all allocated participants. All allocated participants on study received at least 1 dose of study drug.
Groups:
- VARIVAX Adolescents (13 to 17 Years): Participants aged 13 to 17 years of age received 2 doses of VARIVAX™ administered approximately six weeks apart: one 0.5 mL dose of VARIVAX™ administered by SC injection on Day 1, and a second 0.5 mL dose of VARIVAX™ by SC injection on Day 43.
- VARIVAX Children (7 to 12 Years): Participants aged 7 to 12 years of age received one 0.5 mL dose of VARIVAX™ administered by SC injection on Day 1.
- VARIVAX Children (12 Months to 6 Years): Participants aged 12 months to 6 years of age received one 0.5 mL dose of VARIVAX™ administered by SC injection on Day 1.
Arm/Group | VARIVAX Adults (18 to 75 Years) | VARIVAX Adolescents (13 to 17 Years) | VARIVAX Children (7 to 12 Years) | VARIVAX Children (12 Months to 6 Years)
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/30 | 0/33 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/30 | 1/33 | 0/37
Other Adverse Events (participants affected / at risk) | 40/50 | 17/30 | 15/33 | 16/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VARIVAX Adults (18 to 75 Years) (N=50) | VARIVAX Adolescents (13 to 17 Years) (N=30) | VARIVAX Children (7 to 12 Years) (N=33) | VARIVAX Children (12 Months to 6 Years) (N=37)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VARIVAX Adults (18 to 75 Years) (N=50) | VARIVAX Adolescents (13 to 17 Years) (N=30) | VARIVAX Children (7 to 12 Years) (N=33) | VARIVAX Children (12 Months to 6 Years) (N=37)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection site pain (General disorders) | 29 (45) | 10 (14) | 10 (10) | 5 (5)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 5 (5)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 4 (6)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Body temperature increased (Investigations) | 6 (11) | 5 (10) | 2 (2) | 9 (13)
Headache (Nervous system disorders) | 9 (15) | 6 (10) | 5 (5) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 2 (2) | 1 (1)
Injection site erythema (General disorders) | 16 (17) | 1 (1) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 7 (9) | 1 (1) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 3 (6) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will comply with the requirements for publication of study results. In accordance with standard editorial and ethical practice, the Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. If publication activity is not directed by the Sponsor, investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT03843632/Prot_SAP_000.pdf